CLINICAL TRIAL: NCT04014179
Title: A Multi-centre, Practice-level, Cluster Randomized Controlled Trial to Compare Point-of-care HCV RNA Testing, Dried Blood Spot Testing, and Standard of Care to Enhance Treatment Uptake Among People With HCV Who Have Recently Injected Drugs Attending Needle and Syringe Programs: the TEMPO Study
Brief Title: Enhancing Hepatitis C Testing and Treatment Among People Who Inject Drugs Attending Needle and Syringe Programs
Acronym: TEMPO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: VHCRP1904
Record Dates: First submitted 2019-07-07; First posted 2019-07-10 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Hepatitis C; Hepatitis C, Chronic
Keywords: Hepatitis C Virus, Needle and Syringe Programs
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Dried Blood Spot (Intervention) (Experimental): Blood samples will be tested for HCV RNA from dried blood spot cards.
  Interventions: Diagnostic Test: Aptima HCV Quant DX Assay
- Point-of-care RNA (Intervention) (Experimental): Blood samples will be tested for HCV RNA using the Xpert HCV Viral Load Fingerstick point-of-care assay.
  Interventions: Diagnostic Test: Xpert HCV Viral Load Fingerstick
- Standard of Care (Control) (No Intervention): Sites will continue with their standard of care for hepatitis C testing.

INTERVENTIONS:
Diagnostic Test: Xpert HCV Viral Load Fingerstick — The Cepheid Xpert HCV Viral Load (VL) Fingerstick assay is an in vitro nucleic acid amplification test designed for the quantitation of Hepatitis C Virus (HCV) DNA in human whole blood using the automated GeneXpert Systems. The HCV RNA result from the Xpert test will be used to initiate HCV treatment.
  Arms: Point-of-care RNA (Intervention)
Diagnostic Test: Aptima HCV Quant DX Assay — The Aptima HCV Quant Dx assay is a real-time transcription-mediated amplification test.
  The assay is used for both detection and quantitation of hepatitis C virus (HCV) RNA in fresh and frozen human serum and plasma from HCV-infected individuals, and in this study from dried blood spots. The HCV RNA result from the Aptima assay will be used to initiate HCV treatment.
  Arms: Dried Blood Spot (Intervention)

SUMMARY:
This project aims to evaluate two strategies of Hepatitis C virus (HCV) testing compared to standard of care among people who inject drugs at needle and syringe program (NSP) services in Australia, to see if it can improve the number of people who start treatment following an HCV diagnosis:

1. HCV testing from collected dried blood spots sent to a central laboratory
2. HCV testing using a point-of-care device at the NSP site
3. HCV testing using standard of care at the NSP site

DETAILED DESCRIPTION:
The TEMPO study will compare dried blood spot testing and point-of-care HCV RNA testing to standard of care as strategies to enhance HCV treatment uptake among people with HCV and recent injecting drug use attending NSP services. Peer support to enhance engagement and facilitate linkage to nursing care will be provided in the intervention arms of this study.

The study is a cluster randomized controlled trial. The sites (clusters) will be primary NSPs which provide services to people who inject drugs and have capacity to provide hepatitis C treatment services. The sites will be located in Australia.

Eighteen NSPs (the clusters) will be randomly allocated to receive point-of-care HCV RNA testing (6 clusters), dried blood spot testing (6 clusters) or standard of care (6 clusters).

At screening, participants will be tested for HCV infection with dried blood spot, point-of-care or standard of care, depending on cluster randomisation.

Screening will continue until a total of 150 HCV RNA positive participants (~25 participants per site) are enrolled in the dried blood spot arm, 150 HCV RNA positive participants are enrolled in the point-of-care arm, and 150 participants are enrolled in the standard of care arm. Hence a total of 450 HCV RNA positive participants.

HCV RNA negative participants will have no further assessments or visits as part of the study protocol.

Participants who are HCV RNA positive will be enrolled in the follow-up cohort and will be assessed for treatment eligibility. If eligible, they will be treated as per standard of care with a pharmaceutical benefits scheme (PBS) approved pan-genotypic HCV DAA treatment. Participants will be encouraged to take the first dose on the day of treatment work-up where possible. On-treatment and post-treatment testing and monitoring will be based on the site investigator as per standard clinical practice.

All HCV RNA positive participants will be followed up at 12 weeks, 24 weeks and 12 months post enrolment.

ELIGIBILITY:
Inclusion criteria for participants:

Attendees of the NSP service are eligible for inclusion if the following criteria are met:

1. Provided written informed consent
2. ≥ 18 years of age
3. Recent injecting drug use - defined as self-reported use within the previous six months.

Exclusion criteria for participants:

a. Is unable or unwilling to provide informed consent or abide by the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2700 (Estimated)
Dates: Start 2022-07-27 (Actual); Primary Completion 2025-07-22 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of HCV RNA positive who initiate HCV treatment | 12 weeks from Enrolment
  To compare the proportion of HCV RNA positive participants who initiate HCV treatment at 12 weeks following enrolment between those who receive point-of-care HCV RNA testing, dried blood spot testing, and standard of care.

CONTACTS AND LOCATIONS:
Locations (17):
- Australia (17):
  - Bankstown NSP, Bankstown, New South Wales
  - WSLHD Drug Health - Blacktown NSP, Blacktown, New South Wales
  - Coffs Harbour Primary NSP, Coffs Harbour, New South Wales
  - Gosford NSP, Gosford, New South Wales
  - Grafton Primary NSP, Grafton, New South Wales
  - Kempsey Primary NSP, Kempsey, New South Wales
  - Liverpool Southwest NSP, Liverpool, New South Wales
  - WSLHD Drug Health - Mt Druitt NSP, Mount Druitt, New South Wales
  - Orana Centre, Wollongong, New South Wales
  - Alcohol and Drug Harm Reduction Biala, Brisbane, Queensland
  - Severin St NSP (Youth Link), Cairns, Queensland
  - Inala, Inala, Queensland
  - Kobi House, Toowoomba, Queensland
  - UC Adelaide, Adelaide, South Australia
  - Wonggangga Turtpandi Aboriginal Primary Health Care Services, Adelaide, South Australia
  - Northern DASSA, Elizabeth, South Australia
  - Noarlunga Health Precinct, Old Noarlunga, South Australia

IPD SHARING:
Plan to Share IPD: No